CLINICAL TRIAL: NCT04048122
Title: Strategy-based Cognitive Intervention for Parkinson Disease: A Pilot Randomized Controlled Trial
Brief Title: Feasibility and Effect of a Strategy-Based Cognitive Intervention for Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201906062
Record Dates: First submitted 2019-08-01; First posted 2019-08-07 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
Keywords: occupational therapy; cognition
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to treatment arm (1:1 ratio, stratified by sex): the intervention or the standard of care control. Both arms will consist of 10 individualized treatment sessions within a 12-week period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized to treatment arm: the intervention or the standard of care control. Participants will not be informed if their treatment group is the experimental intervention or standard of care.
  Both treatments consist of 10, 1-hour sessions over 12 weeks delivered in an individual, face-to-face format in participants' homes and/or communities by trained licensed occupational therapists (OTs).
  Members of the research team who are involved in the post-treatment testing will be blinded to which intervention (experimental or control) the study participant received from the trained OT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control Group) (Active Comparator): This treatment is task-oriented training, a widely-used approach in neurorehabilitation, that parallels the cognitive process training used in PD to-date but with simulated functional tasks (vs. computer or paper & pencil tasks). It has the same basic protocol as MC4PD, but it is therapist-directed, and the OT does not address strategies, metacognition, generalization, or use mediation or action plans. The OT selects treatment activities based on the client's cognitive profile and goals from a published set of activities designed for use in cognitive interventions. Graded task practice with OT feedback on performance accuracy is used to produce neurocognitive improvement (or possibly independent strategy development). The OT assigns practice of specific cognitively challenging everyday life activities for homework (but without action plans).
  Interventions: Behavioral: Standard of Care
- MC4PD Strategy Training (Experimental): This treatment focuses on improving functional performance by enhancing the generation and use of strategies-which can be internal (e.g., self-talk, planning) or external (e.g., checklist, alarm)-to circumvent cognitive processing limitations caused by PD. It uses a standardized approach across and within sessions for all clients while being tailored to each client's cognitive problems and goals.
  Interventions: Behavioral: MultiContext for PD Strategy Training

INTERVENTIONS:
Behavioral: MultiContext for PD Strategy Training — This treatment is task-oriented training, a widely-used approach in neurorehabilitation, that parallels the cognitive process training used in PD to-date but with simulated functional tasks (vs. computer or paper & pencil tasks). It has the same basic protocol as MC4PD, but it is therapist-directed, and the OT does not address strategies, metacognition, generalization, or use mediation or action plans. The OT selects treatment activities based on the client's cognitive profile and goals from a published set of activities designed for use in cognitive interventions. Graded task practice with OT feedback on performance accuracy is used to produce neurocognitive improvement (or possibly independent strategy development). The OT assigns practice of specific cognitively challenging everyday life activities for homework (but without action plans).
  Arms: MC4PD Strategy Training
Behavioral: Standard of Care — This treatment is task-oriented training, a widely-used approach in neurorehabilitation, that parallels the cognitive process training used in PD to-date but with simulated functional tasks (vs. computer or paper & pencil tasks). It has the same basic protocol as MC4PD, but it is therapist-directed, and the OT does not address strategies, metacognition, generalization, or use mediation or action plans. Therefore, this is a standard-of-care approach that includes all but the proposed critical elements of MC4PD. The OT reviews pre-treatment cognitive test scores with the client but without discussion to build awareness. The OT selects treatment activities based on the client's cognitive profile and goals from a published set of activities designed for use in cognitive interventions.
  Arms: Standard of Care (Control Group)

SUMMARY:
Parkinson disease (PD) affects over 1 million Americans and causes considerable personal and socioeconomic costs (>$34 billion/year in the US) that are expected to rise as the population ages. Cognitive impairment produces disability and reduced quality of life among non-demented people with PD. Surgical and pharmacologic treatments for PD do not prevent or treat cognitive impairment and may even exacerbate the problem. As such, cognitive rehabilitation treatments that mitigate its negative functional consequences are a top research priority.

Unfortunately, existing cognitive rehabilitative programs for PD, which focus on restoring deficient cognitive processes through process training (repetitive practice of tasks that challenge specific cognitive processes), have had limited effect on daily function. To overcome this limitation, the investigators take a strategy training approach. Trained occupational therapists teach people targeted strategies to use in everyday life to circumvent cognitive deficits and accomplish meaningful daily activities. Contemporary cognitive rehabilitation evidence supports this approach for people with chronic neurocognitive dysfunction from stroke and brain injury; however, it has not been studied in PD. By teaching strategies for everyday cognition and using training techniques to support transfer of learning beyond the training context, the investigators hypothesize that our strategy training interventions will produce better functional outcomes for people with PD compared to process training.

The investigators developed MultiContext for PD (MC4PD) to enable people with PD to apply strategies in their everyday lives to cope with cognitive decline and improve or maintain daily function. MC4PD is an individualized, community-based intervention that focuses on the attainment of personally meaningful functional goals using training techniques known to enhance strategy learning and transfer. In an iterative case series, the investigators fine-tuned the treatment protocol, established good participant acceptance and engagement, and provided preliminary data on its benefits for daily cognitive function. The next step is to confirm MC4PD's feasibility in a randomized controlled trial (RCT). In this project, the investigators will assess feasibility and treatment fidelity and generate data in preparation for a definitive RCT by conducting a single-blind pilot RCT comparing MC4PD to a standard-of-care treatment (Control). Individuals with PD will complete pre-treatment testing, randomization to treatment group, 10 treatment sessions, and immediate and 3 months post-treatment testing.

DETAILED DESCRIPTION:
Parkinson disease (PD) affects over 1 million Americans and causes considerable personal and socioeconomic costs (>$34 billion/year in the US) that are expected to rise as the population ages. Cognitive impairment produces disability and reduced quality of life among non-demented people with PD. Surgical and pharmacologic treatments for PD do not prevent or treat cognitive impairment and may even exacerbate the problem. As such, cognitive rehabilitation treatments that mitigate its negative functional consequences are a top research priority.

Unfortunately, existing cognitive rehabilitative programs for PD, which focus on restoring deficient cognitive processes through process training (repetitive practice of tasks that challenge specific cognitive processes), have had limited effect on daily function. To overcome this limitation, the investigators take a strategy training approach. Trained Occupational Therapists teach people targeted strategies to use in everyday life to circumvent cognitive deficits and accomplish meaningful daily activities. Contemporary cognitive rehabilitation evidence supports this approach for people with chronic neurocognitive dysfunction from stroke and brain injury; however, it has not been studied in PD. By teaching strategies for everyday cognition and using training techniques to support transfer of learning beyond the training context, the investigators hypothesize that our strategy training interventions will produce better functional outcomes for people with PD compared to process training.

The investigators developed MultiContext for PD (MC4PD) to enable people with PD to apply strategies in their everyday lives to cope with cognitive decline and improve or maintain daily function. MC4PDis an individualized, community-based intervention that focuses on the attainment of personally meaningful functional goals using training techniques known to enhance strategy learning and transfer. In an iterative case series, the investigators fine-tuned the treatment protocol, established good participant acceptance and engagement, and provided preliminary data on its benefits for daily cognitive function. The next step is to confirm MC4PD's feasibility in a randomized controlled trial (RCT). In this project, the investigators will assess feasibility and treatment fidelity and generate data in preparation for a definitive RCT by conducting a single-blind pilot RCT comparing MC4PD to a standard-of-care treatment (Control). Individuals with PD (N = 60) will complete pre-treatment testing, randomization to treatment group, 10 treatment sessions, and immediate and 3 months post-treatment testing.

Aim 1: Examine the feasibility of MC4PD within an RCT. H1: Study recruitment will be 4 participants/month, retention in both treatment groups will be 4 participants/month, retention in both treatment groups will be > or equal to 85%, and greater than or equal to 85% of participants in both groups will complete the intervention in 12 weeks. The investigators will track recruitment, retention, intervention duration, and reasons for non-enrollment or attrition throughout the study period.

Aim 2: H2a: Therapists will deliver MC4PD with high adherence and competence. Blinded raters will rate therapist adherence and competence for a random sample (30%, n=180) of MC4PD and Control treatment sessions. The investigators will calculate adherence and competence (to MC4PD) for each therapist; adherence > or equal to 80% and competence greater than or equal to 3 (of 4 possible, indicating at least "Well done") will be benchmarks for good treatment integrity. H2b: MC4PD participants will have good acceptance, receipt, and enactment of treatment. MC4PD participants will complete the Client Satisfaction Questionnaire (CSQ-8) at post-treatment, and blinded raters will rate participants' session participation (Pittsburgh Rehabilitation Participation Scale; PRPS) and homework completion. CSQ-8 scores greater than or equal to 24 (of 32 possible, indicating all positive responses), PRPS scores greater than or equal to 4 (of 6, indicating at least "Good"), and homework completion rates greater than or equal to 80% will be benchmarks for good acceptance, receipt, and enactment, respectively.

Aim 3: Obtain preliminary estimates of MC4PD's effect on patient-reported functional cognition. H3 (exploratory): MC4PD participants will report greater improvement in functional cognition than Control participants immediately and 3 months after treatment. The Investigators will use the Bangor Goal Setting Interview (BGSI), a reliable and responsive rehabilitation outcome measure, to identify 3-5 functional cognitive problems and set related goals for each participant. Participants will rate their attainment of each goal at pre, post, and follow-up (10-point scales, higher is better, scores are averaged across problems).

The investigators hypothesize that MC4PD can enable people with PD to manage everyday cognitive challenges so they can perform and participate in desired activities and roles. Such an intervention could improve function and quality of life, reduce caregiver burden, and enhance clinical care for this population. This specific study is part of a rigorous developmental process designed to optimize MC4PD for clinical trials and eventual translation into clinical practice. It is significant because it will provide us with feasibility data, fidelity enhancements, clinical trials infrastructure, experience training and monitoring therapists, and an estimate of treatment effect-all essential elements for efficiency, rigor, reproducibility, and payoff in future clinical trials as well as for implementation and sustainability in real-world clinical practice.

Participants will complete pre-treatment assessment and then will be randomized to treatment arm: MC4PD or Control (Standard of Care). Both arms will consist of 10 individualized treatment sessions within a 12-week period.

Both treatments consist of 10, 1-hour sessions over 12 weeks delivered in an individual, face-to-face format in participants' homes and/or communities by trained licensed occupational therapists (OTs). All treatment sessions will be audiotaped to assess the therapists adherence and competence to the cognitive treatments.

Arm 1 - MC4PD: This treatment focuses on improving functional performance by enhancing the generation and use of strategies-which can be internal (e.g., self-talk, planning) or external (e.g., checklist, alarm)-to circumvent cognitive processing limitations caused by PD. It uses a standardized approach across and within sessions for all clients while being tailored to each client's cognitive problems and goals. The first session begins with a discussion of pre-treatment cognitive test results from the recruitment source study. The purpose of this is to (1) begin building the client's awareness of cognitive strengths and limitations and how they may relate to daily function and (2) inform individualized goal setting and treatment planning. Then the OT explains MC4PD purpose and process, conducts the Bangor Goal Setting Interview to collaboratively identify functional cognitive problems and set related treatment goals, and "assigns" the first homework (record and reflect on daily cognitive lapses). All subsequent treatment sessions consist of a review of prior sessions and learning, homework review, treatment activities, homework provision, and session recap. Each session's treatment activities are selected collaboratively based on the client's goals and preferences and the OT's assessment of the client's cognitive and functional status. They involve the performance of simulated functional activities with OT mediation to help the client anticipate performance problems, generate and use strategies to support performance, evaluate and modify performance and strategy use, and transfer these principles to other activities. The OT's expertise in functional cognition, task and performance analysis, and task grading guides this process. Treatment activities also involve in-depth discussion of these issues, including making explicit connections between the simulated functional activities, strategies, and the client's real-life experiences, to promote generalization of learning. Homework consists of action plans for using the strategies generated and practiced during the treatment session in specific everyday life situations. Clients record instances of strategy use (or missed opportunities) along with their evaluation of strategy effectiveness and potential modifications on a structured worksheet, which is reviewed collaboratively in the next session. In this way, homework not only supports real-life strategy application and practice, but it also reinforces self-monitoring, self-evaluation, problem solving, strategy self-generation, and strategy optimization. Treatment progresses through three general phases (1: Understand and define problems and goals, 2: Generate, execute, and evaluate strategies, 3: Generalize and reinforce strategy use) and increases in difficulty, but progression is flexible depending on the client's goals and abilities.

Arm 2 - Control: This treatment is task-oriented training, a widely-used approach in neurorehabilitation, that parallels the cognitive process training used in PD to-date but with simulated functional tasks (vs. computer or paper & pencil tasks). It has the same basic protocol as MC4PD, but it is therapist-directed, and the OT does not address strategies, metacognition, generalization, or use mediation or action plans. Therefore, this is a standard-of-care approach that includes all but the proposed critical elements of MC4PD. The OT reviews pre-treatment cognitive test scores with the client but without discussion to build awareness. The OT selects treatment activities based on the client's cognitive profile and goals from a published set of activities designed for use in cognitive interventions. Graded task practice with OT feedback on performance accuracy is used to produce neurocognitive improvement (or possibly independent strategy development). The OT assigns practice of specific cognitively challenging everyday life activities for homework (but without action plans).

Participants will complete assessments related to cognition, goal-attainment, participation one-week and three-months post-treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* males and females over age 40 who meet criteria for typical idiopathic PD (stage I-III)
* Have subjective cognitive decline (SCD) as defined by a positive answer to either question: "Do you feel like your thinking skills or memory are becoming worse?" "Do you have problems with your thinking skills or memory?", and can list one or more daily cognitive challenge they wish to address.
* Medications should be stable for 4 weeks prior with no changes planned during the study (we will document unplanned changes).

Exclusion Criteria:

* Dementia according to MDS criteria or a Montreal Cognitive Assessment (MoCA) score < 21
* other neurological disorders
* brain surgery
* history of psychotic disorder
* any condition that would interfere with participation (e.g. non-English speaking, significant current depression)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, Movement Disorders Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foster ER, Carson L, Jonas J, Kang E, Doty T, Toglia J. The Weekly Calendar Planning Activity to Assess Functional Cognition in Parkinson Disease. OTJR (Thorofare N J). 2022 Oct;42(4):315-323. doi: 10.1177/15394492221104075. Epub 2022 Jun 17. PMID 35713209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between November 2019 and January 2022 from the university movement disorders clinic, other research studies, and the community.
Groups:
- Control: This treatment is task-oriented training, a widely-used approach in neurorehabilitation, that parallels the cognitive process training used in PD to-date but with simulated functional tasks (vs. computer or paper & pencil tasks). It has the same basic protocol as MC, but it is therapist-directed, and the OT does not address strategies, metacognition, generalization, or use mediation or action plans. The OT selects treatment activities based on the client's cognitive profile and goals from a published set of activities designed for use in cognitive interventions. Graded task practice with OT feedback on performance accuracy is used to produce neurocognitive improvement (or possibly independent strategy development). The OT assigns practice of specific cognitively challenging everyday life activities for homework (but without action plans).
- Multicontext (MC): This treatment focuses on improving functional performance by enhancing the generation and use of strategies-which can be internal (e.g., self-talk, planning) or external (e.g., checklist, alarm)-to circumvent cognitive processing limitations caused by PD. It uses a standardized approach across and within sessions for all clients while being tailored to each client's cognitive problems and goals. Treatment sessions consist of a review of prior sessions and learning, homework review, treatment activities, homework provision, and session recap. Each session's treatment activities are selected collaboratively based on the client's goals and preferences and the OT's assessment of the client's cognitive and functional status. They involve the performance of simulated functional activities with OT mediation to help the client anticipate performance problems, generate and use strategies to support performance, evaluate and modify performance and strategy use, and transfer these principles to other activities.
Period: Overall Study
Arm/Group | Control | Multicontext (MC)
Started | 28 | 29
Completed | 25 | 26
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Multicontext (MC) | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (7.7) | 71 (6.8) | 70.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 29 | 56
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — A measure of global cognition, with a score range of 0-30 total points, with a higher score indicating better overall cognition.
  units on a scale | 25 (2.7) | 26 (2.2) | 25.5 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bangor Goal Setting Interview (BGSI) Goal Attainment
Description: BGSI is a structured interview schedule was used to record participant ratings of performance and satisfaction in reaching specific goals, and to record additional ratings of goal attainment. This instrument rates goal attainment on a ten point scale (1-10) with a higher score indicating higher goal attainment.
Time Frame: Pre-cognitive treatment intervention; one week post- cognitive treatment intervention (11 to 13 weeks after the pre-cognitive intervention treatment session); and at 3-months follow-up after the post- cognitive treatment treatment session.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Multicontext (MC)
Number analyzed (Participants) | 25 | 26
score on a scale
  Pre-treatment | 4.5 (.3) | 4.6 (.3)
  Post-treatment | 5.9 (.2) | 7.4 (.2)
  Follow-up | 5.6 (.3) | 6.9 (.3)

2. Secondary Outcome: Client Satisfaction Questionnaire
Description: Assesses client satisfaction with intervention provided one week after the cognitive intervention, approximately 11 to 13 weeks). Scores can range from 0 to 32, with a higher score indicating higher satisfaction with the intervention.
Time Frame: Administered one time, one week post- cognitive treatment intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Multicontext (MC)
Number analyzed (Participants) | 25 | 26
score on a scale | 28.8 (3) | 29.3 (3.1)

3. Secondary Outcome: Treatment Fidelity Scale
Description: Measures adherence (1=absent, 2=present) and competence (0=absent, 1=little evidence, 2=adequate/proficient) of the therapist to the MC treatment components (Anticipation, Strategy Generation, Task Challenges, Strategy Post Discussion, Strategy Application). Higher scores are better. This will be completed by a blind rater.
Time Frame: Each of the 10 cognitive treatment intervention sessions. These treatment sessions will be 1 to 1.5 hours in length, and be delivered once a week, to be completed within a 12-week time frame.
Population: A random sample of ~3 treatment sessions per participant.
Measure: Mean (Standard Deviation); unit: Score on fidelity scale
Units Other Than Participants: Treatment sessions
Arm/Group | Standard of Care (Control Group) | MC4PD Strategy Training
Number analyzed (Participants) | 28 | 29
Number analyzed (Treatment sessions) | 67 | 71
Score on fidelity scale
  Anticipation Adherence | 1.0 (0) | 1.8 (.38)
  Strategy Generation Adherence | 1.0 (.03) | 1.8 (.38)
  Task Challenges Adherence | 1.1 (.15) | 1.9 (.29)
  Strategy Post Adherence | 1.1 (.23) | 1.9 (.21)
  Strategy Application Adherence | 1.0 (.10) | 1.9 (.24)
  Anticipation Proficiency | 0 (.03) | 1.5 (.77)
  Strategy Generation Proficiency | 0 (.03) | 1.5 (.75)
  Task Challenges Proficiency | .05 (.15) | 1.7 (.60)
  Strategy Post Proficiency | .09 (.25) | 1.7 (.49)
  Strategy Application Proficiency | .02 (.10) | 1.7 (.47)

ADVERSE EVENTS:
Time Frame: For each participant, from their first treatment session to their post-treatment assessment, so up to 13 weeks. Adverse events were only monitored/ assessed up to their post-treatment assessment.
Description: At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit. In addition, an AE/SAE may occur during a study visit or come to the attention of study personnel in communications with study participants between visits (e.g., calling to cancel an appointment). All events will be captured on the AE/SAE Report Forms.
Arm/Group | Control | Multicontext (MC)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/29
Other Adverse Events (participants affected / at risk) | 8/28 | 15/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=28) | Multicontext (MC) (N=29)
Acute kidney infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Experienced recurrent falls and had OH, so went to the ER; admitted to the hospital for 6 days; determined there was an acute kidney injury/infection that was causing the falls and OH
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=28) | Multicontext (MC) (N=29)
Falls (Musculoskeletal and connective tissue disorders) | 8 (15) | 15 (42) — falls

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT04048122/Prot_SAP_000.pdf